CLINICAL TRIAL: NCT06502197
Title: Comparative Analysis of Short-term (4 Weeks) vs. Long-term (12 Weeks) Silastic Stenting in Frontal Sinus Surgery: A Prospective Study of Clinical Outcomes
Brief Title: Comparative Analysis of Silastic Stenting in Sinus Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Addenbrooke's Hospital, Cambridge University (Unknown); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Arif Janjua, Clinical Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H23-03592
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Chronic Rhinosinusitis, Endoscopic Sinus Surgery, Silastic Stenting
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-term (4 weeks) Silastic Stenting (Experimental)
  Interventions: Procedure: Silastic Stenting
- Long-term (12 weeks) Silastic Stenting (Experimental)
  Interventions: Procedure: Silastic Stenting

INTERVENTIONS:
Procedure: Silastic Stenting — Drill-out frontal sinus procedures, are a well-established surgical intervention in the management of CRS, involves extensive sinus surgery with the creation of a large, surgically exposed area of raw bone. This raw bone, left exposed postoperatively, poses a unique challenge in the context of mucosal healing. Silastic stents, inserted into the sinus cavities, offer a promising solution by providing structural support and facilitating mucosal re-mucolisation in this critical period of postoperative recovery.

SUMMARY:
Silastic stenting is a measure taken to support tissue healing following sinus surgery. Silastic stents are inserted into the sinus cavities and provide structural support while facilitating healing in the critical period of recovery following surgery. There is controversy over the optimal duration for which silastic stents should be left in place. Having them in place for shorter periods may reduce the likelihood of stent-related reactions, while leaving them for longer periods could promote more tissue healing. The aim of this study is to compare the impact of stent duration on clinical outcomes of patients following sinus surgery.

DETAILED DESCRIPTION:
Patients will be recruited consecutively from the PI's frontal sinus surgery list. The research assistant will approach the patient to obtain informed consent before the day of the operation. A written patient information leaflet explaining the study will be provided.

Eligible patients will be categorized into two groups:

* Group A: Short-term stent retention (4 weeks)
* Group B: Long-term stent retention (12 weeks) We aim for a sequence of 50 "4 week-stent" and 50 "12 week-stent". The patients will be told whether they are receiving the stent for 4 or 12 weeks at the day of surgery.

Standard of care:

1. Preoperative visit, assessment including nasal endoscopy and completion of SNOT-22 baseline questionnaire.
2. Surgery with frontal sinus drill out (Draf IIa, IIb, &III) are done as a standard of care in these centers. Dressing of the raw drilled out surface area of the beak with silastic stents is the standard of care for all drill outs.
3. Post-operative follow-ups at 4 weeks and 12 weeks', with 4 weeks vs 12 weeks of stent removal time scale.

Study will require:

1. Categorization of patients into two groups: one group who will have a silastic stent for 4 weeks, and the other group will have stent in place for 12 weeks.
2. Saving a copy of the endoscopic image intra-operative and at 6 months and one-year post-op. To compare the size of a frontal drainage pathway, measuring anterior-posterior & medial-lateral diameters.

Study Process:

At the first pre-operative appointment for drill out, the procedure is discussed. At this point, the study will be introduced by the principal and sub investigators and explained in detail by the research coordinator who would also obtain informed consent. If the patient consents to the study, a SNOT22 (sino-nasal outcome measure 22) pre-operative questionnaire will be completed; thereafter, they will be categorized to one of the two groups.

At time of surgery, frontal stent placement is placed to minimize contracture and to aid with re-mucolisation of the raw surface area due to the drill out, allowing for creation of optimal frontal sinus opening. Therefore, after the maximal desired sinus drill out has been achieved, and the surgeon feels that the surgery proceeded routinely, with no circumstances that would indicate the use of silastic stents for other reasons (such as injury to posterior plate mucosa or 360 mucosal disruption), an envelope that indicates which arm of the study the patient will be opened and the choice for placement of the stent for what time interval would be revealed to the surgeon. In the event of a non-routine surgery, the surgeon will complete the surgery as required by the circumstance, and the patient will be withdrawn from the study. The information about withdrawal will be communicated to the participant immediately post-operative, and during their first routine follow-up appointment.

For all participants that provide informed consent, a routine follow-up endoscopic assessment will be performed as per standard of care at 4 weeks, 12 weeks, 6 months and 1 year. During these examinations an endonasal photograph will be taken for measurement and analyzing. Photographs will be evaluated by two independent surgeons to reduce bias.

At the second and final 1-year postoperative follow-ups, the patients will be asked to complete two brief questionnaires of the patient-reported experience related to healing. Questionnaires on symptoms: one is the validated SNOT22 scoring system and the other was adopted from SNOT22; both address health related issues concerning the quality of life as pertain to sinus disease1. The second questionnaire includes the following items that relate to the study aims:

A) During the post-operative process:

* Nasal obstruction (none-mild-moderate-severe)
* Crusting (none-mild-moderate-severe)
* Cacosmia (none-mild-moderate-severe)
* Halitosis (none-mild-moderate-severe)
* Nasal discomfort (none-mild-moderate-severe)
* Acute sinus infection (when, duration, antibiotic requirement).

B) Experience of the post-operative appointment:

* Pain association with debridement and/or stent removal [graded on a visual analogue scale where 0 is no pain (none) and 10 is the worst (severe) pain ever experienced]
* Did the patients adhere to taken analgesia (Tylenol / Paracetamol) 30 mins pre-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic rhinosinusitis requiring Frontal drill-out.

Exclusion Criteria:

* Patients unwilling or unable to comply with the study protocol.
* Previous Radiotherapy to operated area.

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-02 (Estimated); Primary Completion 2025-09-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Long-Term Patency | 6 and 18 months
  Patency is to be assessed by using the validated scoring system from Lund VJ, Kennedy DW. Quantification for staging sinusitis. In: Kennedy DW, editor. International Conference on Sinus Disease: Terminology, Staging, Therapy. Ann Otol Rhinol Laryngol 1995; 104(Suppl 167):17-21.
Incidence of acute sinus infection | 2 and 4 weeks
  The occurrence and frequency of acute sinusitis in both cohorts, requiring rescue course of oral antibiotics.

SECONDARY OUTCOMES:
Tolerability Assessment | At the respective stent extraction time
  Instrument: Likert Scale
Symptom Relief Assessment | 6 and 18 months post-op
  Instrument: Sinonasal Outcome Test-22 (SNOT-22)